CLINICAL TRIAL: NCT01872026
Title: ASP7991 Clinical Pharmacological Study -Examination of Pharmacokinetics and Pharmacodynamics in Chronic Kidney Disease Patients Undergoing Hemodialysis
Brief Title: Examination of Plasma Concentrations and Safety in Chronic Kidney Disease Patients Undergoing Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 7991-CL-1003
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Patients on Stable Chronic Maintenance Dialysis Who Are Receiving Hemodialysis Therapy; Pharmacodynamics of ASP7991; Pharmacokinetics of ASP7991
Keywords: ASP7991; Plasma concentration; Pharmacodynamics; Pharmacokinetics
MeSH Terms: interventions — ASP7991

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1- single administration (Experimental): The lowest, middle and the highest dose ASP7991 as a single oral administration on non-dialysis day in step 1 to 3 and the highest dose on day of dialysis in step 4.
  Interventions: Drug: ASP7991
- Part 2- repeated administration (Experimental): The lowest, middle and the highest dose ASP7991 as repeated oral administration in step 1 to 3.
  Interventions: Drug: ASP7991

INTERVENTIONS:
Drug: ASP7991 — oral

SUMMARY:
This study is to assess the safety, tolerability, plasma concentration and pharmacodynamics of ASP7991 after oral administration to patients with chronic kidney disease undergoing hemodialysis.

DETAILED DESCRIPTION:
To examine the pharmacokinetics, pharmacodynamics and safety in patients with chronic kidney disease undergoing hemodialysis.

* To assess the pharmacokinetics (PK), pharmacodynamics (PD), safety and the effect of hemodialysis on PK of single oral administration of ASP7991 in Part 1.
* To assess the safety, PK and PD of repeated oral administration of ASP7991 in part 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients on stable chronic maintenance dialysis who are receiving hemodialysis therapy 3 times/week for more than 12 weeks (84 days) and are also scheduled to undergo the regimen of 3 times/week hemodialysis during the study period
* Patients who have secondary hyperparathyroidism;

  1. Receiving Active vitamin D or Cinacalcet hydrochloride
  2. OR iPTH values ≥ 180 pg/mL at screening in case patients receive no medication for secondary hyperparathyroidism.
* Corrected serum Ca at screening：≥ 8.4 mg/dL
* No changes in items below at least 7 days before screening and do not have a plan to change something in the items below during the trial.

  1. Dose and type of Active Vitamin D, Calcitonin preparation, Phosphate binder.
  2. Ca concentration of the dialysate, membrane area of the dialyzer and dialysis time of each week(possible to change within ±10%)

Exclusion Criteria:

* Patients who underwent parathyroid intervention within 24 weeks prior to the informed consent
* Patients who have primary hyperparathyroidism
* Having a history of gastric/intestinal resection considered influential on the absorption of the drug in the gastrointestinal tract
* Patients with uncontrolled hypertension (systolic blood pressure ≥ 180 mmHg and diastolic blood pressure ≥ 120 mmHg are showed at the previous three points at the initiation of dialysis including the screening assessment)
* Complicated by severe heart disorder [congestive cardiac failure (NYHA classification III or higher), or wide range of old myocardial infarction], or having a history of hospitalization for cerebro-vascular disease or heart disorder within 12 weeks(84 days) before obtaining the informed consent.
* Concurrent serious hepatic disease (acute and active chronic hepatitis, hepatic cirrhosis)
* History of malignant tumor
* History of serious drug allergy including anaphylactic shock
* Potentially child-bearing, lactating, those who do not comply with the instructed contraceptive measures
* Patients who were involved in an assessment of other clinical trial within 12 weeks(84 days) prior to the informed consent
* Patients who is an employee of the sponsor, CRO, SMO, or sites related to the study.
* Patients who have been judged ineligible to participate in the study by the investigator / sub investigator.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-12-26 (Actual); Primary Completion 2013-06-26 (Actual); Study Completion 2013-06-26 (Actual)

PRIMARY OUTCOMES:
The safety of ASP7991 assessed by the incidence of adverse events, vital signs, laboratory tests, 12-lead ECGs, ECGs for QT evaluation and ophthalmic examination | For 9-16 days after dosing

SECONDARY OUTCOMES:
Plasma concentrations unchanged drug; AUClast, AUCinf, AUC24h, Cmax, Ctrough, tmax, t1/2, CL/F, Vz/F | For 9-16 days after dosing
iPTH, wPTH, corrected serum Ca* (Serum Ca and Serum Alb), P | For 9-16 days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Kantou, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=276